CLINICAL TRIAL: NCT04886518
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Pitolisant on Excessive Daytime Sleepiness and Other Non-Muscular Symptoms in Patients With Myotonic Dystrophy Type 1, Followed by an Open-Label Extension
Brief Title: Safety and Efficacy of Pitolisant on Excessive Daytime Sleepiness and Other Non-Muscular Symptoms in Patients With Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBS-101-CL-005
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Myotonic Dystrophy 1; Excessive Daytime Sleepiness
MeSH Terms: conditions — Myotonic Dystrophy; Disorders of Excessive Somnolence | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Higher dose pitolisant (Active Comparator): Double-Blind Treatment Phase:
  Week 1: 8.9 mg pitolisant administered once daily in the morning; Week 2: 17.8 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 35.6 mg pitolisant administered once daily in the morning.
  Interventions: Drug: Pitolisant Oral Tablet
- Lower dose pitolisant (Active Comparator): Double-Blind Treatment Phase:
  Week 1: 4.45 mg pitolisant administered once daily in the morning; Week 2: 8.9 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 17.8 mg pitolisant administered once daily in the morning
  Interventions: Drug: Pitolisant Oral Tablet
- Placebo (Placebo Comparator): Double-Blind Treatment Phase:
  Week 1: Matching placebo tablets; Week 2: Matching placebo tablets; Weeks 3 through 11: Matching placebo tablets
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pitolisant Oral Tablet — Pitolisant 4.45 mg tablets: white, round, plain, biconvex film-coated tablet, 3.7 mm in diameter. Each tablet contains 5 mg of pitolisant hydrochloride equivalent to 4.45 mg of pitolisant.
  Pitolisant 17.8 mg tablets: white, round, plain, biconvex film-coated tablet, 7.5 mm in diameter. Each tablet contains 20 mg of pitolisant hydrochloride equivalent to 17.8 mg of pitolisant.
  Arms: Higher dose pitolisant; Lower dose pitolisant
Drug: Placebo oral tablet — Matching placebo tablets will be provided for each strength of active pitolisant film-coated tablets.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of pitolisant compared with placebo in treating excessive daytime sleepiness (EDS) in patients with Myotonic Dystrophy Type 1 ages 18 to 65 years.

The secondary objectives of this study are to assess the impact of pitolisant on fatigue, cognitive function and the burden of disease along with assessing the long-term safety and effectiveness of pitolisant in patients with Myotonic Dystrophy Type 1 ages 18 to 65 years.

DETAILED DESCRIPTION:
The study will consist of a Screening Period, an 11-week Double-Blind Treatment Phase (including a 3-week Titration Period and an 8-week Stable Dose Period), and an optional Open Label Extension (OLE) Phase. The OLE Phase will last approximately one year for each patient or until the Sponsor elects to terminate the study.

Approximately 30 patients ages 18 to 65 years who meet all eligibility criteria will be randomized at the Baseline Visit in a 1:1:1 ratio to lower dose pitolisant, higher dose pitolisant, or matching placebo. In the Double-Blind Treatment Phase, patients will be titrated to their randomized stable dose of study drug during the 3-week Titration Period.

After completion of the 3-week Titration Period, patients will continue to take study drug at their randomized stable dose once daily in the morning upon wakening for an additional 8 weeks of blinded treatment (Stable Dose Period). The duration of the Double-Blind Treatment Phase will be 11 weeks.

Following the 11-week Double-Blind Treatment Phase, eligible patients will be given the opportunity to participate in an optional OLE Phase. During the OLE Phase, all eligible patients will receive treatment with open-label pitolisant. Patients will first undergo a 3-week Titration Period to a maximum target dose, after which they will continue to take their dose of pitolisant once daily in the morning upon wakening until the end of the study. The patient's dose of pitolisant may be adjusted during the OLE phase.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide voluntary, written informed consent.
2. Has a diagnosis of DM1 confirmed by genetic testing (cytosine-thymine-guanine [CTG] repeat of ≥100) from the Screening Visit.
3. Male or female patients ages 18 to 65 years at the time of enrollment.
4. Has a Clinical Global Impression of Severity (CGI-S) assessment of moderate or severe for overall severity of EDS at Screening.
5. If on a wake-promoting treatment that could affect EDS (including stimulants, modafinil, and armodafinil):

   1. Must be on a stable dose for at least 2 months prior to Screening and agree to continue the stable dose for the duration of the Double-Blind Treatment Phase of the study (dose adjustments will be permitted in the OLE Phase).
   2. If not on a stable dose for 2 months prior to Screening, washout for 5 half-lives prior to randomization and agree to remain off these treatments for the duration of the Double-Blind Treatment Phase of the study.
6. Washout of cannabidiol and tetrahydrocannabinol for 28 days prior to randomization and agree to remain off for the duration of the Double-Blind Treatment Phase of the study.
7. Able to walk independently with or without an assistive device (e.g., cane, walker, orthoses allowed).
8. A patient who is a female of child-bearing potential (FCBP) must have a negative serum pregnancy test at the Screening Visit and negative urine pregnancy test at the Baseline Visit and agree to remain abstinent or use an effective method of non-hormonal contraception to prevent pregnancy for the duration of the study and for 21 days after final dose of study drug.
9. In the opinion of the Investigator, the patient is capable of understanding and complying with the protocol and administration of oral study drug.

Exclusion Criteria:

1. Has a diagnosis of another genetic or chromosomal disorder that is distinct from DM1 and that is not being managed adequately in the opinion of the Investigator.
2. Experiences <6 hours on average of sleep per night based on their sleep diary during Screening (patients need to record at least 7 of 10 consecutive nights including 2 nights that fall on a weekend in their sleep diary during Screening).
3. Consistently consumes >600 mg of caffeine per day and is unable/unwilling to reduce caffeine intake to <600 mg per day for the duration of the Double-Blind Treatment Phase of the study; caffeine intake should remain consistent during Screening and throughout the Double-Blind Treatment Phase of the study.
4. Does not agree to discontinue any prohibited medication or substances listed in the protocol.
5. Is currently breastfeeding or planning to breastfeed over the course of the study. Lactating women must agree not to breastfeed for the duration of the study (Double-Blind Treatment Phase and OLE Phase) and for 21 days after final dose of study drug.
6. Participation in an interventional research study involving another investigational medication or device in the 28 days prior to enrollment; patients who undergo a washout of an investigational medication of at least 5 half-lives can be enrolled in the Double-Blind Treatment Phase of the study. Patients considering participation in another interventional research study in the OLE Phase must consult with the Investigator who will consult with the Medical Monitor.
7. Has a primary diagnosis of severe psychiatric illness.
8. Patients taking antidepressants who have not been on a stable dose of their antidepressant for at least 12 weeks prior to Screening; for patients on a stable dose of their antidepressant for at least 12 weeks prior to Screening, must agree to continue their stable dose for the duration of the Double-Blind Treatment Phase of the study. Dose adjustments will be permitted in the OLE Phase. In the Double-Blind Treatment Phase of the study, antidepressants that are strong CYP2D6 inhibitors are exclusionary.
9. Has a history of sleep-disordered breathing or another underlying sleep disorder that in the opinion of the Investigator is a main contributory factor to the patient's EDS.
10. Has a diagnosis of end-stage renal disease (ESRD; estimated glomerular filtration rate [eGFR] of <15 mL/minute/1.73 m2) or severe hepatic impairment (Child-Pugh C).
11. Has a diagnosis of moderate or severe renal impairment (eGFR ≥15 to ≤59 mL/minute/1.73 m2) or moderate hepatic impairment (Child-Pugh B) at Screening or during the Double-Blind Treatment Phase.
12. Has a family history of sudden cardiac death, unexplained death, or death from a primary dysrhythmia potentially associated with QT prolongation in any family member (i.e., first degree relative such as parent, sibling, or offspring).
13. Has a history of unexplained syncope.
14. Has a history of long corrected QT interval (QTc) syndrome or corrected QT interval using Fridericia's formula (QTcF) >450 msec for males or >470 msec for females (QTcF = QT / 3√ RR) sustained atrial fibrillation (AF) or left ventricular ejection fraction <50%.
15. Has a history of documented symptomatic arrhythmias (e.g., ECG, Holter monitor).
16. Electrocardiogram abnormalities during a 10-second, 12-lead ECG at Screening of first degree atrioventricular block (AVB; PR interval >220 msec), QRS >120 msec, heart rate (HR) <50 beats per minute (bpm), marked T-wave abnormalities, more than single atrial premature complexes (APCs) or premature ventricular contractions (PVCs), left bundle branch block, or Brugada pattern type 1.

    Note: Patients with 1st degree AVB with a PR interval >220 msec, who are treated prophylactically with an allowable implanted device are not excluded from the study.
17. Based on Holter monitor, any episode of 3rd degree AVB, any prolonged episode of second degree AVB (>2 episodes during waking hours, >6 episodes during sleep), any prolonged episode of 2nd degree AVB (>10 seconds), any asystole longer than 3.5 seconds, any run of ventricular tachycardia (VT) >6 beats, frequent runs of non-sustained VT (>5/24 hour), >400 PVCs/24 hours, AF or paroxysmal AF, or frequent or complex atrial arrhythmias.
18. Has history of New York Heart Association (NYHA) class III or class IV heart failure.
19. Has an implanted defibrillator or implanted biventricular pacemaker. Note: Patients with implanted univentricular pacemakers that are used prophylactically to prevent or treat bradycardia or heart block may be included.
20. Is receiving a medication known to prolong the QT interval.
21. Has a history of clinically significant hypokalemia or hypomagnesemia that cannot be adequately controlled by supplementation.
22. Has serum potassium or magnesium levels that are outside of the normal reference ranges and considered clinically significant at Screening. Patients with mild hyperkalemia that, in the opinion of the Investigator, does not pose an arrhythmia threat may be included.
23. Is receiving a concomitant medication that is known to be a strong cytochrome P450 (CYP) 2D6 inhibitor, a strong CYP3A4 inducer; or a centrally acting histamine 1 receptor (H1R) antagonist (sedating antihistamine).

    Note: Patients who undergo a washout of these medications of at least 5 half-lives may be enrolled in the Double-Blind Treatment Phase of the study.

    Note: Use of strong CYP2D6 inhibitors and strong CYP3A4 inducers is allowed during the OLE Phase; however, adjustment of pitolisant dose is required. Although not prohibited during the OLE Phase of the study, use of centrally acting or sedating H1R antagonists should be avoided.
24. Is a known CYP2D6 poor metabolizer (PM).
25. Regular use (more than twice per week) of any sleep-promoting treatments that could affect EDS and not willing to limit use to no more than twice per week during Screening and for the duration of the Double-Blind Treatment Phase of the study (use of sleep-promoting agents are not allowed within one day prior to study-related assessments).
26. Has abnormal laboratory values at Screening that are clinically significant as determined by the Investigator.
27. Has initiated any new or change in allied health therapies or interventions that can interfere with the study outcomes within 28 days prior to randomization and that are prohibited during the Double-Blind Treatment Phase of the study, based on the Investigator's judgment.
28. Has a current or recent (within 1 year) history of a substance use disorder or dependence disorder, including alcohol and caffeine use disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V).
29. Has planned surgery during the Double-Blind Treatment Phase of the study; planned surgery is permitted during the OLE Phase.
30. Has a significant risk of committing suicide or suicidality based on history, routine psychiatric examination, Investigator's judgment, or who has an answer of "yes" on any question other than questions 1 to 3 on the Columbia-Suicide Severity Rating Scale.
31. Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to an unstable or uncontrolled medical condition or one that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the patient, or compromise the integrity of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - UCI Center for Clinical Research, Irvine, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Kennedy Krieger Institute Center for Genetic Muscle Disorders, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Hôpital de Chicoutimi, Chicoutimi, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Ambrosio ES, Chuang K, David WS, Amato AA, Gonzalez-Perez P. Frequency and type of cancers in myotonic dystrophy: A retrospective cross-sectional study. Muscle Nerve. 2023 Aug;68(2):142-148. doi: 10.1002/mus.27801. Epub 2023 Mar 27. PMID 36790141

RESULTS

PARTICIPANT FLOW:
Groups:
- Higher Dose Pitolisant: Pitolisant 35.6 mg administered once daily in the morning upon wakening
- Lower Dose Pitolisant: Pitolisant 17.8 mg administered once daily in the morning upon wakening
- Placebo: Matching placebo administered once daily in the morning upon wakening
Period: Overall Study
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Started | 10 | 10 | 10
Completed | 8 | 9 | 10
Not Completed | 2 | 1 | 0
Not completed — Noncompliance with study drug | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 36.5 [20 to 55] | 42.0 [28 to 50] | 41.0 [27 to 60] | 40.0 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 10 | 10 | 29
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 5 | 3 | 12
  United States | 6 | 5 | 7 | 18
Daytime Sleepiness Scale (DSS) [Mean (Standard Deviation); unit: units on a scale] — The score of the Daytime Sleepiness Scale (DSS) ranges from 0 to 15. The higher the score, the higher the degree of daytime sleepiness. Population: The analysis population for this study-specific baseline measure is the modified Intent-to-Treat Population, which includes 8 participants in the higher-dose pitolisant group, 8 in the lower-dose pitolisant group, and 9 in the placebo group.
  units on a scale
    number analyzed (Participants) | 8 | 8 | 9 | 25
    (all) | 8.5 (3.21) | 7.3 (1.16) | 7.9 (3.22) | 7.8 (2.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Excessive Daytime Sleepiness (EDS) Based on Change in Daytime Sleepiness Scale (DSS) Score
Description: The score of the DSS ranges from 0 to 15. A decrease in the DSS score represents an improvement in EDS.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline DSS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 8 | 9
score on a scale | -3.8 (1.98) | -1.8 (1.91) | 0.0 (2.29)

2. Secondary Outcome: Change in Fatigue Based on Change in Fatigue Severity Scale (FSS) Score
Description: The score of the FSS ranges from 0 to 63. A decrease in the FSS score represents an improvement in fatigue.
Time Frame: Baseline to Week 11
Population: The analysis population includes all randomized participants who received at least one dose of study drug and have on baseline and at least one post-baseline FSS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 9 | 10
score on a scale | -0.86 (1.487) | -0.36 (0.367) | -0.13 (0.529)

3. Secondary Outcome: Change in Psychomotor Function Based on Change in Cogstate Detection Test
Description: The Cogstate Detection Test is a computerized test. A faster speed represents an improvement in psychomotor test performance.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline Cogstate assessment.
Measure: Mean (Standard Deviation); unit: log10 ms
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7 | 8
log10 ms | 0.02 (0.058) | -0.05 (0.061) | 0.01 (0.037)

4. Secondary Outcome: Change in Attention Based on Change in Cogstate Identification Test
Description: The Cogstate Identification Test is a computerized test. A faster speed represents an improvement in attention test performance.
Time Frame: Baseline to Week 11
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 ms
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7 | 8
log10 ms | 0.00 (0.035) | -0.02 (0.076) | -0.02 (0.052)

5. Secondary Outcome: Change in Working Memory Based on Change in Cogstate One Back Test
Description: The Cogstate One Back Test is a computerized test. A faster speed represents a better working memory test performance.
Time Frame: Baseline to Week 11
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 ms
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 7 | 6 | 8
log10 ms | 0.00 (0.062) | -0.01 (0.032) | 0.00 (0.050)

6. Secondary Outcome: Change in Burden of Disease Based on Change in Myotonic Dystrophy Health Index (MDHI)
Description: The MDHI score ranges from 0 to 100. A decrease in the MDHI score represents an improvement in overall burden of disease.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline MDHI assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 9 | 10
score on a scale | -9.14 (13.277) | -2.89 (8.510) | 0.42 (5.529)

7. Secondary Outcome: Change in Excessive Daytime Sleepiness (EDS) Based on Change in Epworth Sleepiness Scale (ESS) Score
Description: The score of the ESS ranges from 0 to 24. A decrease in the ESS score represents an improvement in EDS.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline ESS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 9 | 10
score on a scale | -4.9 (3.98) | 1.3 (2.83) | -0.1 (2.51)

8. Secondary Outcome: Change in Excessive Daytime Sleepiness (EDS) Based on Change in Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S is a one-item scale that ranges from 0 to 4 with 0 being no EDS and 4 being severe EDS. The scale is completed by the site investigator/clinician. The higher the CGI-S score, the more severe the clinician's perception of the patient's symptoms of EDS.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline CGI-S assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 9 | 10
score on a scale | -0.9 (0.64) | -0.2 (0.44) | -0.1 (0.32)

9. Secondary Outcome: Change in Excessive Daytime Sleepiness (EDS) Based on Change in Patient Global Impression of Severity (PGI-S)
Description: PGI-S is a one-item scale that ranges from 0 to 4 with 0 being no EDS and 4 being severe EDS. The scale is completed by the patient. The higher the PGI-S score, the more severe the patient's perception of excessive daytime sleepiness.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline PGI-S assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 8 | 9 | 10
score on a scale | -0.5 (0.76) | 0.0 (1.0) | -0.4 (0.84)

10. Secondary Outcome: Change in Sustained Attention Based on Sustained Attention to Response Task (SART)
Description: The Sustained Attention to Response Test provides a measure of vigilance and sustained attention. A number ranging from 1 to 9 is presented on screen. The subject must press a predetermined button (the YES external button) as soon as the number is presented, except when the number is a 3. The number 3 is the default number (no-go stimulus) for which a response should be inhibited, and the subject should not press the predetermined button. The no-go stimulus can be configured to be a number other than 3. Performance is measured by calculating the number of errors made during the test over the course of 225 trials. Performance is measured by calculating the error score, which is the sum of trials where a response was provided when a 3 was presented and trials where no response was provided when a number other than 3 was presented.
  A decrease in the SART score represents an improvement in sustained attention.
Time Frame: Baseline to Week 11
Population: This analysis population includes all randomized participants who received at least one dose of study drug and have one baseline and at least one post-baseline Sustained Attention to Response Task assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
Number analyzed (Participants) | 6 | 7 | 8
scores on a scale | -2.33 (5.428) | 1.43 (4.467) | 21.88 (68.689)

ADVERSE EVENTS:
Time Frame: Data presented for adverse events occurring from the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 11 weeks.
Description: The Double-Blind safety population included all patients who were enrolled and took at least one dose of double-blind study drug.
Groups:
- Higher Dose Pitolisant: Pitolisant 35.6 mg administered once daily in the morning
- Lower Dose Pitolisant: Pitolisant 17.8 mg administered once daily in the morning
- Placebo: Matching placebo administered once daily in the morning
Arm/Group | Higher Dose Pitolisant | Lower Dose Pitolisant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose Pitolisant (N=10) | Lower Dose Pitolisant (N=10) | Placebo (N=10)
Headache (Nervous system disorders) | 5 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 4 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Migraine (Nervous system disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thirst decreased (General disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04886518/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04886518/SAP_001.pdf